CLINICAL TRIAL: NCT02849249
Title: A Prospective, Multicenter, Randomized, Controlled, Open Trial, Parallel Groups (1: 1), With Subcutaneous Polimerized Mix (100/100), in Patients With Rhinoconjunctivitis Sensitized to the Following Combination of Pollen: Timothy Grass and Olea Europaea, and Asministered by Different Schedules
Brief Title: A Trial With Subcutaneous Immunotherapy (SCIT) in Patients With Rhinoconjunctivitis Sensitized to Olea Europaea and Phleum Pratense
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roxall Medicina España S.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIA-OLEAPHL-POLI-100
Record Dates: First submitted 2016-07-22; First posted 2016-07-29 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Rhinoconjuntivitis
Keywords: allergy; Immunotherapy; SCIT
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- One day schedule (Active Comparator): Allergovac polimerized with a mixture of 2 pollen extracts (100:100): Olea europea and Phleum pratense, administered in one day schedule. The maintenance dose (0.5 mL) is reached in one day.
  Interventions: Biological: allergovac polimerized (100/100)
- Rapid schedule (Active Comparator): Allergovac polimerized with a mixture of 2 pollen extracts (100:100): Olea europea and Phleum pratense, administered in a rapid Schedule.The initation phase includes 3 weekly increasing doses till the maintenance dose of 0.5 mL is reached.
  Interventions: Biological: allergovac polimerized (100/100)

INTERVENTIONS:
Biological: allergovac polimerized (100/100) — Patients will recieve a initiation phase plus a mantenaince phase for 3 months of an allergy vaccine.
  Other Names: Allergovac Poliplus

SUMMARY:
The study was designed according to the draft of allergenic product regulation published by Spanish Regulatory Agency. The aim of the study is to evaluate the safety and tolerability of subcutaneous immunotherapy with polimerized (100/100) mixture of pollens: Olea europaea and Phleum pratense in patients with rhinoconjunctivitis with or without associated mild asthma. In addition, surrogate efficacy parameters will be evaluated: immunoglobulin level changes and skin reactivity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must sign the Informed Consent Form.
2. Patients must be between 18 and 60 years of age.
3. Patients with seasonal allergic rhinoconjunctivitis produced by Phleum pratense and Olea europaea during at least 2 years prior to participating in the study. Although the pathology being studied is allergic rhinoconjunctivitis, patients who have concomitant mild or moderate asthma may be included.
4. Patients who have had a skin prick test result ≥ 3 mm in diameter against Phleum pratense and Olea europaea.
5. Patients who have specific IgE ≥ class 2 (CAP/PHADIA) to Phleum pratense and Olea europaea.
6. Patients will preferably be polysensitized to Phleum pratense. Polysensitized patients to otherallergenic sources may only be included in the study if their other sensitizations are produced by:

   1. Overlapping seasonal pollens which are cross-reactive with Phleum pratense and Olea europaea.
   2. Pollens whose seasons do not overlap with Phleum pratense or Olea europaea and which are not expected to produce symptoms during the study period.
   3. Other allergens which are not expected to produce symptoms during the study period.
7. Women of child-bearing potential must have a negative urine pregnancy test at the time they begin the study.
8. Furthermore, women of child-bearing potential must agree to use adequate contraceptive methods during this study if they are sexually active.

Exclusion Criteria:

1. Patients who received immunotherapy in the previous 5 years for Phleum pratense and Olea europaea or for any allergen with cross reactivity or patients that are currently receiving immunotherapy for any allergen.
2. Patients with severe asthma or forzed expiratoy volumen in 1 second FEV1< 70% even if the are pharmacologically controlled .
3. Patients with: immunological, cardiac, renal or hepatic illnesses or any other medical condition that the investigator deems relevant so as to interfere with the study.
4. Patients with a previous history of anaphylaxis
5. Patients with chronic urticaria,
6. Patients with moderate to severe atopic dermatitis
7. Patients who have participated in another clinical trial within 3 month prior to enrolment.
8. Patients under treatment with tricyclic antidepressives, phenothiazines , β- blockers, or Angiotensin Converting Enzyme Inhibitors (ACEI)
9. Female patients who are pregnant or breast-feeding
10. Patient who does not attend the visits

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number and severity of adverse reactions as a measure of safety and tolerabitity | Across 12-15 weeks treatment period

SECONDARY OUTCOMES:
Immunoglobulin changes from baseline | At baseline and 1 week after last administered dose
  Subrogate efficacy
Skin reactivity changes from baseline | At baseline and 1 week after last administered dose
  Subrogate efficacy parameter. The patients will undergo a skin prick test at baseline and 1 week after last administered dose. The wheal are in mm2 will be measured and the results of both time frames will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: María C Gómez, Dr., Study Director — Roxall Medicina España S.A
Locations (5):
- Spain (5):
  - Hospital de Zafra, Zafra, Badajoz
  - Hospital de Henares, Henares, Madrid
  - Hospital Clínico Granada, Granada
  - Hospital Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville